CLINICAL TRIAL: NCT04532073
Title: Sub-study of the Essen Study Centre With Proteome and Telomer Analyses and Qualitative Parameters for the ENTAiER Trial
Brief Title: Sub-study of the Essen Study Centre for the ENTAiER Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Software AG Stiftung (Unknown); Universität Freiburg (Unknown)
Responsible Party: Principal Investigator, Holger Cramer, Research Director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-9421-BO
Record Dates: First submitted 2020-08-20; First posted 2020-08-31 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Elderly Patients; Chronically Ill; Increased Risk of Falling
MeSH Terms: conditions — Chronic Disease | interventions — Tai Ji; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eurythmy therapy exercises (Experimental): As part of the ENTAiER trial: In group sessions á 5 patients with a qualified therapist: In the first 3 months twice a week, in the second 3 months once a week. Recommendation to practice at home on at least 3 days per week (optimal, practice daily). They are supported by an eurythmy manual and an exercise video. This supplements the regular care.
  Interventions: Other: Eurythmy Therapy
- Tai Chi exercises (Experimental): As part of the ENTAiER trial:In group sessions of 5 patients each with a qualified teacher: In the first 3 months twice a week, in the second 3 months once a week. Recommendation to practice at home on at least 3 days per week (optimal, practice daily). They are supported by a Tai Chi Manual and an exercise video. This complements the regular care
  Interventions: Other: Tai Chi
- Standard Care Only (Active Comparator): As part of the ENTAiER trial:Brochure with detailed description of various evidence-based measures for fall prevention, prepared for the specific age group (https://www.trittsicher.org/files/trittsicher_bzga_sturzpraevention_2015-11-23.pdf)
  - Recommendation to visit the family doctor and discuss fall prophylaxis with her
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Eurythmy Therapy — A mindfulness-oriented movement therapy
  Arms: Eurythmy therapy exercises
Other: Tai Chi — A martial art developed in China, which in recent times is often regarded as a system of movement theory or gymnastics
  Arms: Tai Chi exercises
Other: Standard Care — Treatment process that a clinician should follow for a certain type of patient
  Arms: Standard Care Only

SUMMARY:
The present study is a sub-study of the ENTAiER study. The ENTAiER study is a multicenter, randomized, controlled study to evaluate the efficacy and safety of eurythmy therapy and Tai Chi in comparison to standard care in chronically ill older patients with an increased risk of falling.

In addition to the main questions of the ENTAiER study, three additional questions are being investigated at the Hospital Essen-Steele: Proteome and telomere analyses as well as qualitative parameters are recorded and examined. The aim is to compare the changes in proteomes, telomeres and qualitative factors under eurythmy therapy, Tai Chi and standard care in chronically ill older patients with an increased risk of falling.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years.
* Chronic disease (musculoskeletal, neurological, internal medicine).
* Increased risk of falling (Berg Balance Scale Score 49 or less).
* Medical history: feeling of balance disturbance in the past.
* Independent living at home or in an old people's or retirement home.
* Regular participation in a one-hour event is possible.
* Sufficiently mobile to leave the place of residence independently at least twice a week
* Written declaration of consent.

Exclusion Criteria:

* Disease that restricts participation (e.g. terminal disease, heart failure NYHA III-IV, unstable angina pectoris, uncontrolled seizure disorder, decompensated lung disease that already leads to shortness of breath during light activity, advanced cancer, chemo- or radiotherapy ongoing or during the last 3 months, amputation of one or both legs)
* Complete dependence on the rollator.
* Visual, hearing or speech problems that limit the understanding of the study documents and processes.
* Major cognitive impairment (MoCA score 18 or less).
* High risk of needing individual supervision during group sessions.
* Severe personality disorder or psychiatric illness, alcoholism or other substance dependence affecting the group sessions.
* Life expectancy under 1 year.
* Permanent bed-riddenness expected in less than one year.
* Regular participation in Tai Chi or EYT in the last 6 months.
* Participation in intensive sports activities in the last month (e.g. training in the fitness centre or in sports groups which lead to breathlessness and sweating; skiing, mountaineering in high mountains).
* Patients who cannot understand the nature, meaning and necessities of participating in a study.
* Participation in another clinical trial within 3 months prior to screening for the ENTAiER trial or concurrent participation in another trial that may interfere with this trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change in proteomic analysis from baseline to after intervention | Before intervention (week 0) and after intervention (6 months)
  A maximum of 500 µL plasma is used for the proteomic studies. The proteins are digested tryptically, a concentration determination is performed by amino acid analysis and the peptide samples are then measured by different mass spectrometric methods (data dependent (DDA) and independent detection (DIA), proteome-wide prediction of peptide tandem mass spectra by deep learning (Prosit), etc.). The results obtained are then verified by Western blot, ELISA and/or a targeted mass spectrometric method (parallel reaction monitoring)
Change in telomer analysis from baseline to after intervention | Before intervention (week 0) and after intervention (6 months)
  The telomere length is determined from blood samples using quantitative real-time PCR (TaqMan) from genomic DNA.
Qualitative parameter | After intervention (6 months)
  By means of semi-structured interviews of maximum 60 minutes per participant, the effects of the intervention are to be recorded qualitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Main study — https://www.drks.de/drks_web/navigate.do?navigationId=trial.HTML&TRIAL_ID=DRKS00016609